CLINICAL TRIAL: NCT00187447
Title: Comparison of 2 Different Indomethacin Dosing Protocols to Treat Infants Delivered at <28 Weeks Gestation With a Persistent Patent Ductus Arteriosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: RC1
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2005-09

CONDITIONS: Patent Ductus Arteriosus
Keywords: prematurity; chronic lung disease; necrotizing enterocolitis; indomethacin; ductus arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth; Enterocolitis, Necrotizing | interventions — Indomethacin

INTERVENTIONS:
Drug: indomethacin (two different dosing regimens)

SUMMARY:
The purpose of this study is to examine if a higher dose of indomethacin will increase the rate of ductus arteriosus closure in extremely premature infants without increasing the side effects. The long term objective is to find the optimal dosing of indomethacin for permanent closure of the Ductus and prevent the morbidity related to PDA and the complications of surgical ligation.

DETAILED DESCRIPTION:
This study is a Phase II randomized, masked, controlled trial that compares the current standard dose of indomethacin to a higher dose for the closure of PDA in premature infants less than 28 weeks of gestation.

Neonates (<28 weeks gestation) who are started on indomethacin treatment (with an initial 3-dose course: 0.2, 0.1, and 0.1 mg/kg of indomethacin) within the first 96 hr after birth will be eligible for this trial if they continue to have Doppler evidence of ductus patency before the third dose of indomethacin. This group of infants have greater than 65% chance of developing symptomatic PDA and surgical ligation even after our standard extended course of indomethacin. Those infants who do not fit the exclusion criteria will be randomized to either a Standard Dose group or to a Higher Dose group after obtaining consent. The infants randomized to the standard group will receive a 4th, 5th, and 6th dose of indomethacin (0.1 mg/kg) at 24 hr intervals (starting at 24 hr after the 3rd dose). The Higher Dose group infants delivered between 26-27 weeks gestation will receive a 4th, 5th, 6th, 7th, 8th and 9th dose of indomethacin (0.1mg/kg) at 12 hr intervals (starting 12 hr after the 3rd dose). The Higher Dose group infants between 24-25 weeks gestation will receive a 4th, 5th, 6th, 7th, 8th and 9th dose of indomethacin (0.25mg/kg) at 12 hour intervals (starting 12 hr after the 3rd dose). To keep the study blinded, the standard group will receive 3 extra doses of saline to match the 3 additional doses given to the higher dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn infants of less than 28 weeks gestational age who are treated with indomethacin during the first 48 hours after birth
2. Presence of patent ductus arteriosus (PDA) by Doppler echocardiography between the second and third dose of indomethacin.
3. Creatinine ≤1.8 mg/dl
4. Platelets ≥ 50,000

Exclusion Criteria:

1. Chromosomal disorders.
2. Major congenital anomalies.
3. Contraindications for indomethacin

   1. Necrotizing enterocolitis, by clinical or radiological evidence
   2. Evidence of bleeding diathesis as evidenced by pulmonary hemorrhage, persistent oozing from puncture sites, grossly bloody stool (Note: Infants with an intracranial hemorrhage can be enrolled in this study).

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2003-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The incidence of ductus closure, as determined by echocardiography, following the last dose of study drug
The incidence of the appearance of a symptomatic PDA following the last dose of study drug
The incidence of ductus ligation.

SECONDARY OUTCOMES:
Altered renal function during treatment
Incidence of Necrotizing enterocolitis
Incidence of chronic lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Clyman, M.D., Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California San Francisco, Davis, California
  - University of Chicago, Chicago, Illinois
  - Brown University, Providence, Rhode Island